CLINICAL TRIAL: NCT01545713
Title: A Phase II, Prospective, Single-center Study: Correlation of Donor-specific Anti-precursor Endothelial Cells With Transplant Outcome for Recipients of Living-donor Kidney Transplants, Are Auto-antibodies Important.
Brief Title: Correlation of Donor-specific Anti-endothelial Cells
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Friedewald, Associate Professor of Medicine and Surgery, Northwestern University
Other Study IDs: XM-One AbSorber
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Living-Donor Kidney Transplants
Keywords: renal; kidney; transplant; living donor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A total of 40 cc/3 tablespoons of blood will be drawn once.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Transplant Recipients: Patients undergoing living-donor kidney transplant at NMH who have a positive XM-One AbSorber® positive test result.

SUMMARY:
Antibody Mediated Rejection (AMR) is a major complication of solid organ transplantation. The main reason for AMR is pre-formed, or de-novo, donor specific antibodies against the donor human leukocyte antigens (HLA). Additional potential targets are antibodies against MIC-A antigens or antibodies against targets expressed on the donor endothelial cells.

Until recently, no specific means were available to test for the presence of donor-specific endothelial cell antibodies. The newly introduced XM-One AbSorber® assay allows isolating precursor endothelial cells from donor peripheral blood, and thus assessing the presence of donor-specific endothelial cell antibodies.

XM-One AbSorber® is an in-vitro assay that allows for the specific enrichment of precursor endothelial cells which in turn promotes endothelial cells specific cross match testing.

This assay is currently being used in an on-going Northwestern University (NU) research study (STU#00029988). The preliminary results of this study indicate that indeed some of the patients test positive against their respective donors. One potential explanation for this observation, that was not previously entertained, is that the antibodies causing the positive cross match response are actually of autoimmune nature. In order to rule-out such a potential explanation the investigators would like to further test these patients by performing an autologous XM-One AbSorber® assay in which the recipient sera will be incubated with the patients' own cells (as opposed to the respective donor cells in the parental study). This information is crucial for proper analysis of the data obtained in the NU STU#00029988 study.

DETAILED DESCRIPTION:
Antibody Mediated Rejection (AMR) is a major complication of solid organ transplantation. The main reason for AMR is pre-formed, or de-novo, donor specific antibodies against the donor HLA antigens. Additional potential targets are antibodies against MIC-A antigens or antibodies against targets expressed on the donor endothelial cells.

Until recently, no specific means were available to test for the presence of donor-specific endothelial cell antibodies. The newly introduced XM-One AbSorber® assay allows isolating precursor endothelial cells from donor peripheral blood, and thus assessing the presence of donor-specific endothelial cell antibodies.

XM-One AbSorber® is an in-vitro assay that allows for the specific enrichment of precursor endothelial cells which in turn promotes endothelial cells specific cross match testing.

This assay is currently being used in an on-going Northwestern University (NU) research study (STU#00029988). The preliminary results of this study indicate that indeed some of the patients test positive against their respective donors. One potential explanation for this observation, that was not previously entertained, is that the antibodies causing the positive cross match response are actually of autoimmune nature. In order to rule-out such a potential explanation we would like to further test these patients by performing an autologous XM-One AbSorber® assay in which the recipient sera will be incubated with the patients' own cells (as opposed to the respective donor cells in the parental study). This information is crucial for proper analysis of the data obtained in the NU STU#00029988 study.

Initial data from our laboratory indicates that the antigens identified by the XM-One Absorber® assay differ from the HLA antigens usually identified by routine cross match assays. Moreover, we were able to document that this is a polymorphic system and therefore identifying a donor-specific source is critical.

Of the 150 patients already studied under NU research protocol STU#00029988 we found that 19 patients exhibited a positive response in a donor-specific XM-One AbSorber® assay. In this current research protocol study we want to follow-up on the specimens that exhibited a positive response in a donor-specific XM-One AbSorber® assay and perform an autologous XM-One AbSorber® assay to validate the clinical significance of our results.

There has been one multicenter study reported indicating the "XM-One AbSorber® is a quick, easy to perform on whole blood samples and identifies patients at risk for rejection and reduced graft function not identified by conventional lymphocyte cross matches" The primary objective is to complete additional testing for accuracy to determine whether antibodies directed at donor-specific endothelial cell effect transplant outcome.

The secondary objective is to assess the frequency of autologous antibodies that may be falsely reported as donor-specific anti-endothelial antibodies in our patient population. The single center research study we here at Northwestern University have been working on since May 19, 2010 thus far has resulted in 19 out of 150 specimens tested, have positive results based on the XM-One AbSorber® assay.

In this prospective study we plan to include all XM-One AbSorber® positive test results from all recipients of living-donor kidney transplants performed at Northwestern Memorial Hospital (NMH) since May 19, 2010 initial Institutional Review Board (IRB) approval until 250 transplants are performed. For this research protocol we will be targeting patients to consent only these individuals who have received a XM-One AbSorber® positive test result.

Each donor / recipient pair are required to send peripheral blood samples to the HLA laboratory prior to the scheduled transplant in order to perform lymphocyte cross match (to detect donor specific HLA antibodies; this is (SOC) standard of care). Left over serum and cells from these tests are being used to isolate an enriched precursor endothelial cell population and perform the XM-One AbSorber® assay (NU research protocol #STU00029988).

XM-One AbSorber® assay results - both autologous and allogeneic - will be captured and compared with graft outcome measurements at 3, 6, and 12 months post-transplant. Transplant outcome will be recorded as creatinine levels at the specific time points, protocol and for-cause biopsy results within the first year post transplant, diagnosis of acute cellular or humoral rejection, variation in immunosuppression levels, and any other complications.

Patients that exhibit a positive XM-One AbSorber® allogeneic cross match result will be requested to donate 4 green top tubes of peripheral blood. Cells obtained from this blood will be used in an autologous XM-One AbSorber® cross match assay using the original serum sample used for the allogeneic XM-One AbSorber® cross match assay.

ELIGIBILITY:
Inclusion Criteria:

1. patients older than 18 years of age
2. patients undergoing living-donor kidney transplant at NMH who have a positive XM-One AbSorber® positive test result

Exclusion Criteria:

1. patients undergoing deceased donor kidney transplant
2. patients younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living-Donor kidney transplant recipients at Northwestern Memorial Hospital 18 year of age or older.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To complete additional testing for accuracy | June 2011 - February 2012
  The primary objective is to complete additional testing for accuracy to determine whether antibodies directed at donor-specific endothelial cell effect transplant outcome.

SECONDARY OUTCOMES:
To assess the frequency of autologous antibodies. | June 2011 - February 2012
  To assess the frequency of autologous antibodies that may be falsely reported as donor-specific anti-endothelial antibodies in our patient population. The single center research study we here at Northwestern University have been working on since May 19, 2010 thus far has resulted in 19 out of 150 specimens tested, have positive results based on the XM-One AbSorber® assay.

CONTACTS AND LOCATIONS:
Overall Officials: John Friedewald, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States